CLINICAL TRIAL: NCT06425744
Title: The Effect of Self-Myofascial Release and Pilates Reformer Exercise on Pain, Muscle Function and Quality of Life in Women With Chronic Low Back Pain
Brief Title: Impact of Pilates and Myofascial Release on Women's Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahmyook University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYU 2022-07-014
Record Dates: First submitted 2024-05-10; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Low Back Pain
Keywords: low back pain; Pilates; Myofasical Release; Pain; Flexibility
MeSH Terms: conditions — Low Back Pain; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental 1 group (Active Comparator): The experimental 1 group perform self-myofascial release and Pilates exercises.
  Interventions: Other: self-myofascial release combined reformer Pilates
- experimental 2 group (Active Comparator): The experimental 2 group perform pilates exercise using reformer.
  Interventions: Other: Reformer Pilates

INTERVENTIONS:
Other: self-myofascial release combined reformer Pilates — The self-myofascial release combined reformer Pilates group performs 10 minutes of self-myofascial release using the BALLance© method before beginning 20 minutes of Reformer Pilates. The 6-week program includes warm-up and breathing, main supine exercises 1 and 2, and movements targeting the sacroiliac and hip joints.
  All Pilates exercises are designed in a variety of positions including supine, prone, sitting and standing. All participants attend twice a week for 6 weeks, for a total of 12 sessions.
  And all participants performed home exercise program follows the guidelines of Geroge et al (2021) and includes myofascial release and Pilates Reformer exercises, as well as stretching exercises beneficial for chronic low back pain. The home exercises are performed three times a week for 15 minutes, and exercise materials are distributed.
  Arms: experimental 1 group
Other: Reformer Pilates — The reformer Pilates group will do 30 minutes of Pilates on the Reformer. All Pilates exercises are designed in a variety of positions including supine, prone, sitting and standing. All participants also attend twice a week for 6 weeks, for a total of 12 sessions.
  The home exercise program follows the guidelines of Geroge et al (2021) as well as stretching exercises beneficial for chronic low back pain. The home exercises are performed three times a week for 15 minutes, and exercise materials are distributed.
  Arms: experimental 2 group

SUMMARY:
The aim of this study is to find out if Reformer Pilates and self-myofascial release are effective for pain and muscle function in women with chronic low back pain. Investigators will also look at changes in quality of life. The main questions for the study are

Can Reformer Pilates and self-myofascial release reduce pain in participants? Can Reformer Pilates and self-myofascial release change muscle function in participants? The researchers want to compare the effects of Reformer Pilates and self-myofascial release in women with chronic low back pain.

Participants will be

Group 1 Perform Reformer Pilates and self-myofascial release exercises twice a week for 6 weeks, for a total of 12 sessions.

Group 2 Perform Reformer Pilates exercises twice a week for 6 weeks, for a total of 12 sessions.

Participants will visit the Pilates Centre for an examination before and once after starting the programme.

All groups perform a home exercise training programme for 15 minutes three times a week.

ELIGIBILITY:
Inclusion Criteria:

* People who have had chronic low back pain for 12 weeks or more
* Have a Korean Oswestry Disability Index (KODI) score of 17% or higher

Exclusion Criteria:

* Patients with low back pain due to trauma, neurological lesions of the lower extremities, herniated disc lesions, hip, pelvic or abdominal surgery
* Patients who have received radiation or injections within the last 3 months,
* Pregnant women or patients who have given birth within the last year

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-11-05 (Actual)

PRIMARY OUTCOMES:
Pain severity | From enrollment to the end of treatment at 6 weeks
  Pain severity is measured using a visual analogue scale, where participants mark the level of back pain they feel on a line between 0 mm and 100 mm(0: no pain, 10: worst pain imaginable).
  Measurement unit is in mm, with higher scores considered more painful
Functional disability caused by low back pain | From enrollment to the end of treatment at 6 weeks
  The Korean version of the Oswestry Disability Index (KODI) is used to assess functional impairment due to low back pain. This assessment consists of 10 items, including pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sexual life, social life, and travel, with each item scored on a scale of 0 to 5 for a total of 50 points. The KODI score is given as a percentage (%) of the total score. Scores are categorised as mild disability (0-20%), moderate disability (21-40%), severe disability (40-60%) and disability affecting all aspects of life (>60%), with high test-retest reliability (r=0.92).

SECONDARY OUTCOMES:
Flexibility of lower back and hamstring | From enrollment to the end of treatment at 6 weeks
  Flexibility is measured using the sit-to-stand reach test (SRT), which assesses the flexibility of the lower back and hamstrings. The score is the most distant point (cm) reached with the fingertips. The best of three trials should be recorded. Participants sit with their feet on a box, knees straight, and reach as far forward as possible. The posture is maintained for five seconds and the reach distance is recorded over three trials and averaged. The longer the distance in centimeters, the more flexible it is.
Muscular endurance | From enrollment to the end of treatment at 6 weeks
  Muscular endurance is assessed using the supine bridge test (SBT), which requires participants to raise their pelvis to form a straight line from shoulder to knee. The time taken to hold the position is recorded in seconds (sec) and averaged over three trials. The longer time hold is the higher muscular endurance.
Quality of life questionnaire | From enrollment to the end of treatment at 6 weeks
  The European Quality of Life 5-Dimensional 5-Level Version (EQ-5D-5L) questionnaire is used to assess quality of life. This standardised tool assesses five dimensions: mobility, self-care, activities of daily living, pain/discomfort, and anxiety/depression. General health status is measured using a visual analogue scale (EQ-5D VAS). Scores on the EQ-5D index range from -0.59 to 1, with 1 being the best health. In the absence of a scoring algorithm, a summed scale score was also calculated for both versions to provide additional information about the contribution of the two additional 5L response categories.

CONTACTS AND LOCATIONS:
Locations (1):
- Pilates Dasom, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No
only IPD used in the results publication